CLINICAL TRIAL: NCT00716326
Title: The Use of Transcutaneous Electrical Nerve Stimulation (TENS) for Chronic Pain of Predominantly Peripheral Neuropathic Origin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8589 (REK); 15602 (NSD); 408/06-301.0 (Fondet)
Record Dates: First submitted 2008-07-09; First posted 2008-07-16 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Neuropathic Pain
Keywords: Transcutaneous Electrical Nerve Stimulation; Chronic pain; Neuropathic pain; Short-term efficacy; Long-term efficacy
MeSH Terms: conditions — Neuralgia; Chronic Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Subjects in this study arm will receive active treatment with Cefar TENS device which delivers therapeutic electrical currents 2-3x over sensory threshold in the area of pain.
  Interventions: Device: Transcutaneous Nerve Stimulation (TENS); Device: Cefar Primo Pro TENS device
- 2 (Placebo Comparator): Subjects in this study arm will receive placebo treatment with manipulated Cefar TENS device which delivers electrical currents just below sensory threshold in the area of pain.
  Interventions: Device: Cefar Primo Pro TENS device

INTERVENTIONS:
Device: Transcutaneous Nerve Stimulation (TENS) — Patients will be randomly allocated to a group with active-TENS and exercises, or to a group with placebo-TENS and exercises. The TENS will be used during 3-4 weeks of hospitalization. If patients want to continue the use of TENS/placebo-TENS at home, they will be offered to borrow equipment for 4 months.
  Arms: 1
Device: Cefar Primo Pro TENS device — Patients will be randomly allocated to a group with active-TENS and exercises, or to a group with placebo-TENS and exercises.
  Active TENS: high-frequency modulated pulse duration stimulation Placebo TENS: manipulated device with impulses near sensory threshold.

SUMMARY:
The aim of this study is to investigate the effectiveness of TENS in addition to routine care in patients with chronic pain of predominantly neuropathic origin, compared to treatment with routine care alone."

Hypothesis:

An eventually neuropathic pain component is needed to be identified and alleviated in chronic pain patients to improve the quality of rehabilitation.

0-hypothesis:

* TENS is not better than than placebo, medication or standard rehabilitation program.
* A neuropathic pain component does not demand special considerations in rehabilitation of chronic pain patients.

DETAILED DESCRIPTION:
Setting:

Skogli helse- og rehabiliteringssenter, Lillehammer, Norway. Center of Rehabilitation for chronic pain patients, rheumatic diseases and orthopedic postoperative patients.

Duration:

Until 18 months of intervention + 6 months of follow up and preparation.

Intervention:

Use of TENS during 3-4 weeks of hospitalization connected to multimodal rehabilitation (short-term efficacy). TENS or placebo-TENS is added to routine care.

Follow-up:

If patients want to continue the use of TENS/placebo-TENS at home, they will be offered to borrow equipment for 4 months. Questionnaires will be send at 2 and 4 months, both for the active group, the placebo group and for the group of patients who discontinued the use of TENS/placebo-TENS (long-term efficacy).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with chronic pain of predominantly neuropathic origin

Exclusion Criteria:

* Pain less than 3 months
* Surgery or lesion within 3 months
* Central neuropathic pain
* Fibromyalgia
* Primary headaches
* Primary psychiatric diagnosis
* Patients with pacemaker
* Formerly treated with TENS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Reduction of pain and/or functional improvement | 3-4 weeks, 2 and 4 months

SECONDARY OUTCOMES:
Compliance. Patient global impression of change | 3-4 weeks, 2 and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan M Bjordal, professor, Study Director — University of Bergen
Locations (1):
- Skogli helse- og rehabiliteringssenter, Lillehammer, Lillehammer, Norway